CLINICAL TRIAL: NCT07026812
Title: Impact of Screens on Children's Growth
Acronym: ECROIPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/138/OB; ID RCB : 2021-A01115-36 (Other: ANSM)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-01

CONDITIONS: Growth Disorders
Keywords: Growth hormone
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Growth hormone stimulation test group

SUMMARY:
Short stature is defined as a height less than -2 Standard Deviations (SD) for age and a slowing of growth velocity by a loss of 1 SD/year. The causes of short stature are multiple (chronic diseases, growth hormone deficiency, hypothyroidism, hyperadrenocorticism, genetic syndromes, etc.). However, nearly 30% are considered idiopathic, with no identified etiology (Naccache et al., unpublished).

Growth hormone (GH) is secreted in a pulsatile manner with maximum peaks primarily at night, raising questions about the relationship between sleep disturbances and short stature.

In children, one of the main causes of sleep disturbances in the digital age is screen use, which is becoming increasingly important, particularly in the pediatric population.

DETAILED DESCRIPTION:
During the night, physiologically, the retina, which no longer receives light signals, sends a message to the suprachiasmatic nucleus, the main key element of the internal clock, and to the pineal gland, which synthesizes melatonin, the sleep hormone. Exposing screens to blue light therefore disrupts melatonin secretion, which leads to a disruption of the circadian rhythm and therefore sleep. Note that this effect of light on melatonin secretion depends on the time of day of exposure, the intensity, and the duration. Thus, exposure to screens before bedtime can be responsible for a delay or even an absence of melatonin synthesis, particularly in the case of nighttime awakenings.

While many studies have examined the impact of screens on children's psychological balance, weight, etc., none, to our knowledge, has examined the potential impact of screens on children's height growth. Hypothesis of this project: 70% of GH synthesis takes place at night, a few minutes after entering slow-wave sleep, sleep disturbed by screens could mean a lower secretion of GH and consequently a delay in height growth.

The objective of this project is to evaluate the impact of screen consumption on sleep and the impact of sleep on idiopathic growth disorder.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 16 years old coming to the day hospital for a growth hormone stimulation test or an oral provocation test (without growth disorders)
* Not opposed to participating in the study
* Patients affiliated with the Social Security system

Exclusion Criteria:

* Growth hormone deficiency confirmed by 2 tests
* Hypothyroidism
* Hypercorticism
* All chronic diseases
* Skeletal pathologies: Turner syndrome, constitutional bone disease Intrauterine growth retardation
* Pubertal delay defined by absence of puberty onset >13 years in girls and 14 years in boys
* Patient under guardianship

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any patient coming to the day hospital for a growth hormone stimulation test and/or for an oral provocation test in the context of an allergy,
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Screen consumption on sleep | At enrollment visit
  Evaluation of the Impact of Screen Consumption on Sleep by Answers to the Questionnaire Given to the Child and/or Parent(s) (Depending on Age)
Screen consumption on sleep | At enrollment visit
  Sleep assessment by responses to the questionnaire given to the child and/or the parent(s) (depending on age) in order to assess the duration of sleep
Screen consumption on sleep | At enrollment visit
  Evaluation of the Impact of Screen Consumption on Sleep by Answers to the Questionnaire Given to the Child and/or Parent(s) (Depending on Age) in Order to Evaluate child's physical activity
Impact of sleep on idiopathic growth disorder | At enrollment visit
  Collection of auxological data at the time of the day hospital consultation (height) noted in the health record and/or in the hospital medical file
Impact of sleep on idiopathic growth disorder | At enrollment visit
  Collection of auxological data at the time of the day hospital consultation (weight) noted in the health record and/or in the hospital medical file
Impact of sleep on idiopathic growth disorder | At enrollment visit
  Collection of auxological data at the time of the day hospital consultation (age) noted in the health record and/or in the hospital medical file

SECONDARY OUTCOMES:
Impact of screens on body size (BMI) | At enrollment visit
  Evaluation of the impact of screens on body size (BMI) by response to the questionnaire given to the child and/or the parent(s)

CONTACTS AND LOCATIONS:
Overall Officials: Mireille MC CASTANET, Professor, Principal Investigator — University Hospital, Rouen; Mireille MC CASTANET, Professor, Study Director — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.